CLINICAL TRIAL: NCT00225641
Title: COLOFOL - A Pragmatic Study to Assess the Frequency of Surveillance Tests After Curative Resection in Patients With Stage II and III Colorectal Cancer - a Randomised Multicentre Trial
Brief Title: Assessment of Frequency of Surveillance After Curative Resection in Patients With Stage II and III Colorectal Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Bispebjerg Hospital (Other)
Collaborators: Nordic Cancer Union (Other); Danish Cancer Society (Other); Danish Colorectal Cancer Group (Unknown)
Responsible Party: Principal Investigator, Peer Wille-Jørgensen, Peer Wille-Jørgensen, DMSc, Bispebjerg Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COLOFOL; Danish Cancer Union 56 100 306
Record Dates: First submitted 2005-09-22; First posted 2005-09-26 (Estimated); Last update posted 2015-12-22 (Estimated); Status verified 2015-12

CONDITIONS: Colorectal Cancer
Keywords: Follow-up
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 frequent control (Active Comparator): Follow-up 6, 12, 18, 24 and 36 months after surgery
  Interventions: Procedure: CT-scan, CEA, X-ray of lungs
- 2 less frequent control (Other): Follow-up 12 and 36 months after surgery
  Interventions: Procedure: CT-scan, CEA, X-ray of lungs

INTERVENTIONS:
Procedure: CT-scan, CEA, X-ray of lungs — Arm 1: 6, 12, 18, 24 and 36 months after surgery
  Arms: 1 frequent control
Procedure: CT-scan, CEA, X-ray of lungs — Arm 2: 12 and 36 months after surgery
  Arms: 2 less frequent control

SUMMARY:
The aim is to conduct a prospective multicentre randomised study comparing two different control regimens after resection for colorectal cancer stage II - III. Follow-up after surgery for colorectal cancer is a controversial issue. The reasons for follow-up are: to obtain a better overall survival, for scientific purposes and/or for psychological reasons and/or as quality assessment. Meta-analyses of randomised controlled studies have lately shown that a beneficial effect on the overall mortality could be found with intense follow-up compared to sporadic. This study compares the regimen of CT-scan or MR scan of the liver, control of the carcinoembryonic antigen (CEA), and CT-scan or X-ray of the lungs in two groups with either control after 12 and 36 months, or after 6, 12, 18, 24, and 36 months. The efficacy parameters are total and cancer-specific mortality.

DETAILED DESCRIPTION:
The aim is to investigate the efficiency of two follow-up programs after radical surgery for colorectal cancer. Colorectal cancer attacks between 3-5% of the European population during their lifetime, and about 75% of these will have potential curative surgery performed. Follow up after surgery is costly and time consuming for both patients and the Health Care Systems. The intensity of follow up as well as the methods employed vary tremendously from center to centre and from country to country. Until recently the scientific documentation for the cost-effectiveness of follow-up was very sparse, but recent compiling of data indicates that intense follow up can save lives as compared to sporadic follow-up at an acceptable cost. However, the optimal follow-up intervals and the best methods are unknown. Previous results indicate that scanning of the liver and measuring of the tumor-marker CEA may be a way forward. A prospective randomised multicenter study in centers from Denmark (approx. 15), Sweden (approx. 20), Poland (approx. 6), Hungary (approx. 2) and perhaps The Netherlands and UK is starting in 2005 after basic work with protocols, ethical committees now has been finished. This basic work was supported by the Nordic Cancer Union with a grant of 25,000 EUROS. The patients will be randomised to follow-up with CEA, multislice CT scan of the liver and X-ray of the lungs, either 12 and 36 months after surgery or 6, 12, 18, 24 and 36 months after surgery. If recurrence is detected, the patient will be offered the best available treatment either as repeated surgery with curative intent or palliative oncological treatment. Data will be collected electronically via the internet to an already constructed database. The primary efficacy parameter is 3 and 5 years overall and cancer-specific survival. It is planned that recruitment will be at least 2,500 patients, which is feasible in 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Radical surgery (R0-resection) for colorectal adenocarcinoma - with or without adjuvant treatment
* Age < 75 years
* Provision of written informed consent for participation
* "Clean colon" verified by perioperative barium enema or colonoscopy last 3 months post-surgery
* Tumour stage: II-III (Tany N1-2 M0, T3-4NanyM0, Dukes´ B - C)

Exclusion Criteria:

* A clinical diagnosis of HNPCC (non hereditary polyposis colorectal cancer) or FAP (familial polyposis coli)
* Local resection for colorectal cancer (e.g., TEM-procedure)
* Life-expectancy less than 2 years due to concurrent disease (e.g., cardiac disease, terminal multiple sclerosis, liver cirrhosis)
* Inability to provide informed consent or refusal to do so
* Inability to comply with the control or intense follow-up program
* Participation in other clinical trials interfering with the control-programs
* Previous malignancies (except for non-melanoma skin cancer)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2500 (Estimated)
Dates: Start 2006-03; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Overall and cancer-specific mortality | 5 years

SECONDARY OUTCOMES:
Quality of life. Cost-effectiveness of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Peer Wille-Jørgensen, Ass Prof., Principal Investigator — Bispebjerg Hospital, Denmark; Adam Dziki, Principal Investigator — Medical University of Lodz, Poland; Nils Lundqvist, Principal Investigator — Norrtälje Hospital, Sweden; Michael Goldinger, Principal Investigator — St.Görans Hospital, Stockholm, Sweden; Mats Bragmark, Principal Investigator — Danderyd Hospital, Stockholm, Sweden; Ulrik Lindforss, MD Phd, Principal Investigator — Södertälje Hospital, Sweden; Kennet Smedh, Principal Investigator — Central Hospital, Västerås, Sweden; Monika Svanfeldt, Principal Investigator — Karolinska University Hospital; Johan Ottoson, Principal Investigator — Central Hospital, Kristianstad, Sweden; Anna Martling, Principal Investigator — Karolinska University Hospital, Solna, Sweden; Jonas Bengtson, Principal Investigator — Sahlgrenska University Hospital; Birger Sandzén, Principal Investigator — University Hospital of Umeå, Sweden; Ingvar Syk, Principal Investigator — Malmö Academic Hospital, Sweden; Lars Påhlman, Principal Investigator — Uppsala University Academic Hospital, Sweden; Pamela Buchwald, Principal Investigator — Helsingborg Hospital, Sweden; Erling Østergaard, Principal Investigator — Viborg Hospital, Denmark; Per Andersen, Principal Investigator — Fyn Hospital, Svendborg, Denmark; Mogens Madsen, Principal Investigator — Herning Hospital, Denmark; Karl Erik Jensen, Principal Investigator — Esbjerg Hospital, Denmark; Per Gandrup, Principal Investigator — Aalborg Hospital, Denmark; Per Jess, Principal Investigator — Hillerød hospital, Denmark; Henrik Christensen, Principal Investigator — Aarhus Hospital, Denmark; Luis Carriquiry, Principal Investigator — Maciel Hospital, Montevideo, Uruguay; Jósef Kladny, Principal Investigator — Pomeranian Medical University, Poland; Christoffer Odensten, Principal Investigator — Sunderby Hospital, Luleå, Sweden; Yngve Raab, Principal Investigator — Södersjukhuset, Stockholm, Sweden; Allan G Pedersen, Principal Investigator — Randers Hospital, Denmark; Helena Laurell, Principal Investigator — Mora Hospital, Sweden; Ronan O'Connel, Principal Investigator — St. Vincents Hospital, Dublin, Ireland
Locations (1):
- Peer Wille-Jørgensen, Copenhagen, Denmark

REFERENCES:
- [Derived] Sorensen HT, Horvath-Puho E, Petersen SH, Wille-Jorgensen P, Syk I; COLOFOL Study Group. More vs Less Frequent Follow-Up Testing and 10-Year Mortality in Patients With Stage II or III Colorectal Cancer: Secondary Analysis of the COLOFOL Randomized Clinical Trial. JAMA Netw Open. 2024 Nov 4;7(11):e2446243. doi: 10.1001/jamanetworkopen.2024.46243. PMID 39570590
- [Derived] Wille-Jorgensen P, Syk I, Smedh K, Laurberg S, Nielsen DT, Petersen SH, Renehan AG, Horvath-Puho E, Pahlman L, Sorensen HT; COLOFOL Study Group. Effect of More vs Less Frequent Follow-up Testing on Overall and Colorectal Cancer-Specific Mortality in Patients With Stage II or III Colorectal Cancer: The COLOFOL Randomized Clinical Trial. JAMA. 2018 May 22;319(20):2095-2103. doi: 10.1001/jama.2018.5623. PMID 29800179